CLINICAL TRIAL: NCT04429399
Title: Effects of Positive End Expiratory Pressure (PEEP) Decrease in Patient With Acute Respiratory Distress Syndrome (ARDS) Ventilated According to High PEEP Strategy (ExPress Trial).
Brief Title: Lowering PEEP: Weaning From High PEEP Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Salvatore Grasso, Associate Professor, University of Bari
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 6011
Record Dates: First submitted 2020-06-04; First posted 2020-06-12 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High positive end-expiratory pressure Ventilation (Other): patient ventilated fixing high level of positive end expiratory pressure
  Interventions: Other: decrease the positive end expiratory pressure (PEEP); Other: mechanical features assessment; Other: shunt assessment
- Low positive end-expiratory pressure Ventilation (Other): patient ventilated fixing low level of positive end expiratory pressure
  Interventions: Other: mechanical features assessment; Other: shunt assessment

INTERVENTIONS:
Other: decrease the positive end expiratory pressure (PEEP) — decrease the PEEP going from high (according to ExPress Trial) to low level
  Arms: High positive end-expiratory pressure Ventilation
Other: mechanical features assessment — evaluation of the mechanical features of respiratory system
Other: shunt assessment — evaluation of the pulmonary shunt during two different ventilation setting

SUMMARY:
The perfusion of the deeply different areas coexisting in ARDS lung generates two type of venus-admixure : true shunt and shunt effect. Briefly, true shunt and shunt effect are related to non-aerated and poorly-ventilated lung areas perfusion respectively. Practically, it is not possible to quantify the true shunt and the shunt-effect directly, but we can measure the "total-shunt", i.e. the sum of two kind of venus-admixured. As it is known from classical physiology, the effects of FiO2 variations on PaO2 are deeply different depending on the type of venous admixures. In the case of a patient with virtually only true shunt, any FiO2 variation will not modify the PaO2. On the other hand, in a patient with virtually only a shunt effect, increasing the FiO2 the PaO2 will progressively increase. Indeed, ventilating a patient presenting only a shunt effect (without true shunt) with pure oxygen will generate a "normal" P/F ratio. In patients ventilated with high PEEP levels it is difficult to predict based on the P/F ratio the relative amount of true shunt and shunt effect. However, patients presenting a significant shunt effect when ventilated with higher PEEP level would likely have "unstable" poorly aerated lung areas that need PEEP to remain opened. In those patients, a PEEP-weaning protocol based on the P/F ratio could induce significant alveolar de-recruitment and clinical deterioration. On the contrary, patients with less shunt effect would be likely less prone to alveolar de-recruitment and would benefice from PEEP decrease.

DETAILED DESCRIPTION:
the investigators set up a study to test the hypothesis that patients presenting a significant shunt effect when ventilated with higher PEEP levels could be prone to significant alveolar de-recruitment at the PEEP weaning attempt. To do so, the investigator has to measure the total shunt at higher PEEP level in patients ready to be weaned from the PEEP (according to the Mercat protocol), at three FiO2 levels (i.e. 0,3, 0,6 and 1). The shunt effect is quantified as the difference in total shunt between FiO2 0,3 and .The hypothesis of this study is that the shunt effect could predict alveolar de-recruitment when weaning PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Age major than 18
* 1-2 days since the beginning of mechanical ventilation
* Moderate or severe ARDS

Exclusion Criteria:

* Patients with a story of chronic obstructive pulmonary disease (COPD)
* Patients with asthma
* Patients with neurological disease
* Patients with heart disease
* Patients with cardiopulmonary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
de-recruitment | decreasing PEEP from high to low levelthrough study completion, an average of 2 years
  the shunt effect cold predict the lung de-recruitment volume

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico, Bari, Italy